CLINICAL TRIAL: NCT05485870
Title: Early Screening and Identification for Panvascular Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021YFC2500502
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Panvascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, feces, urine, saliva, tissue samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Panvascular disease group: patients with panvascular diseases
- Healthy controls: Healthy controls

SUMMARY:
Identify the pathogenic factors involved in the occurrence and development of panvascular disease and its pathogenesis.

DETAILED DESCRIPTION:
Identify the pathogenic factors involved in the occurrence and development of panvascular disease and its pathogenesis by a multi-omics study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with panvascular diseases; 2. Patients or guardians who agreed to join the study; 3. Patients who can complete the relevant examinations involved in this study;

Exclusion Criteria:

* patients with coagulation dysfunction.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with panvascular diseases
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Any new stroke events | Up to 48 months
  Incidence of any new ischemic or hemorrhagic stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No